CLINICAL TRIAL: NCT05705466
Title: A Two-Part, Phase 1b/2, Multicenter, Open-Label, Dose Escalation and Double-Blind, Randomized, Placebo-Controlled, Dose Expansion Study of the Safety, Efficacy and Pharmacokinetics of Navtemadlin Plus Pembrolizumab as Maintenance Therapy in Subjects With Locally Advanced and Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of Navtemadlin Plus Pembrolizumab as Maintenance Therapy in Locally Advanced and Metastatic Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KRT-232-119
Record Dates: First submitted 2023-01-17; First posted 2023-01-30 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Navtemadlin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Navtemadlin in combination with pembrolizumab (Experimental): Navtemadlin will be administered orally, once daily (QD), on days 1-7 in a 21-day cycle.
  Pembrolizumab will be administered intravenously on Day 1 of a 21-day cycle.
  Interventions: Drug: Navtemadlin; Drug: Pembrolizumab
- Navtemadlin placebo in combination with pembrolizumab (Placebo Comparator): Navtemadlin placebo will be administered orally, once daily (QD), on days 1-7 in a 21-day cycle.
  Pembrolizumab will be administered intravenously on Day 1 of a 21-day cycle.
  Interventions: Drug: Navtemadlin Placebo; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Navtemadlin — Navtemadlin is an experimental MDM2 anticancer drug taken by mouth.
  Other Names: KRT-232
  Arms: Navtemadlin in combination with pembrolizumab
Drug: Navtemadlin Placebo — Navtemadlin placebo is a placebo that is the same in appearance to navtemadlin drug taken by mouth.
  Arms: Navtemadlin placebo in combination with pembrolizumab
Drug: Pembrolizumab — Pembrolizumab is a humanized antibody used in cancer immunotherapy that will be administered intravenously
  Other Names: Keytruda

SUMMARY:
This study evaluates Navtemadlin (KRT-232) in combination with Pembrolizumab as a maintenance therapy in patients with locally advanced and metastatic non small cell lung cancer.

DETAILED DESCRIPTION:
This is a 2 part, phase 1b/2, maintenance study for patients who have achieved a partial response (PR) or complete response (CR) after completion of up to 4 cycles of a combination platinum-based chemotherapy plus CPI regimen.

Phase 1b is a 3+3 dose escalation design that will be used to determine the maximum tolerated dose (MTD) and/or the recommended phase 2 dose (RP2D) of navtemadlin in combination with pembrolizumab. A Safety Review Committee (SRC) will review the safety data during the dose escalation to decide on dose escalation and/or exploration of intermediate doses.

Phase 2 will evaluate the efficacy and safety of the RP2D of navtemadlin plus pembrolizumab compared to navtemadlin placebo plus pembrolizumab. Each Arm will have approximately 40 subjects enrolled for a total of approximately 80 subjects. Eligible subjects will be randomized 1:1. This part of the study has a randomized, controlled, double-blind design. A stratified, permuted-block randomization scheme will be used for treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-1
* Histologically or cytologically confirmed diagnosis of NSCLC documented as TP53WT
* Locally advanced or metastatic disease; must have completed up to 4 cycles of platinum-based chemo plus CPI and achieved a CR or PR per RECIST V1.1
* Adequate hematologic, hepatic and renal function (within 14 days)

Exclusion Criteria:

* Symptomatic or uncontrolled central nervous system (CNS) metastases
* Prior treatment with a MDM2 inhibitor
* Grade 2 or higher QTc prolongation (>480 msec per NCI-CTCAE criteria version 5.0)
* History of bleeding diathesis; major hemorrhage or intracranial hemorrhage within 24 weeks
* History of major organ transplant
* Active pneumonitis or known history of interstitial lung disease, drug-related pneumonitis, or radiation pneumonitis
* Prior radiotherapy, cytoreductive therapy, cytokine therapy or any investigational therapy within 28 days
* Medical condition, serious intercurrent illness, psychiatric condition or other circumstance that, in the Investigator's judgment could jeopardize the subject's safety, or that could interfere with study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1b- To determine the recommended Phase 2 dose (RP2D) | 21 days
  The Safety Review Committee will determine the RP2D based on safety data of the combination of navtemadlin and pembrolizumab.
Phase 2- To assess the treatment effect of navtemadlin plus pembrolizumab treatment on PFS compared with the treatment effect of navtemadlin placebo plus pembrolizumab treatment. | 64 Months
  PFS is defined as the time from randomization date to disease progression (assessed by the Independent Review Committee [IRC] per RECIST v1.1) or death, whichever occurs first

SECONDARY OUTCOMES:
Phase 1b- To characterize the pharmacokinetic (PK) profile of navtemadlin | 1 day
  Will determine the Maximum observed concentration (Cmax) on Cycle 1 Day 1
Phase 1b- To characterize the pharmacokinetic (PK) profile of navtemadlin | 1 day
  Will determine the area under the plasma concentration versus time curve (AUC) on Cycle 1 Day 1
Phase 1b- To characterize the pharmacokinetic (PK) profile of navtemadlin | 1 day
  Will determine the time of maximum plasma concentration (Tmax) on Cycle 1 Day 1
Phase 1b- To assess the treatment effect on progression-free survival (PFS) | 64 Months
  PFS is defined as the time from first dose date to disease progression (assessed by the IRC and Investigator per RECIST v1.1) or death, whichever occurs first
Phase 2- To assess the treatment effect of navtemadlin plus pembrolizumab treatment on PFS compared with the treatment effect of navtemadlin placebo plus pembrolizumab treatment. | 64 Months
  PFS is defined as the time from randomization date to disease progression (assessed by the Investigator per RECIST v1.1) or death, whichever occurs first